CLINICAL TRIAL: NCT06725472
Title: Comparison of the Classic Median Sternotomy Skin Incision with the Paramedian Flap Skin Incision Technique in Open Heart Surgery
Brief Title: Comparison of the Classical Median Sternotomy Skin Incision with the Paramedian Flap Skin Incision
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Eyüpserhat ÇALIK, Associate Professor, Ataturk University
Other Study IDs: TSA-2023-13179
Record Dates: First submitted 2024-07-20; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-07

CONDITIONS: Surgical Incision; Surgical Site Infection; Keloid Scar Following Surgery
Keywords: open heart surgery; median sternotomy; flap skin incision
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Paramedian flap skin incision group: Patients undergoing open heart surgery with median sternotomy undergo a skin incision 2-3 cm lateral to the sternum's medium.
  Interventions: Procedure: Open Heart Surgery
- Control group: Patients undergoing open heart surgery with median sternotomy undergo a classical skin incision on the medium of the sternum.
  Interventions: Procedure: Open Heart Surgery

INTERVENTIONS:
Procedure: Open Heart Surgery — This is a general term for surgical procedures that directly access the heart through an opening in the chest to treat heart problems.

SUMMARY:
The goal of this observational study is to determine the effects of a flap-shaped paramedian skin incision on protection from mediastinal infections, wound healing, and scar formation in open heart surgery performed through the classic median sternotomy approach compared with the classic median skin incision. The main question aimed to be answered is:

Is paramedian flap skin incision effective in improving sternotomy wound healing? Does it have a preventive effect on the development of sternal wound infection? Does it have a protective effect on keloid formation? Patients who underwent open-heart surgery with classical median sternotomy will be randomized into two groups: paramedian flap skin incision and median skin incision. The effectiveness of the paramedian incision will be investigated by comparing perioperative data and data from the first three months of follow-up.

DETAILED DESCRIPTION:
Median sternotomy (MS) is the classic opening technique for open heart surgery. The skin incision is made in line with the bone incision at the center of the sternum. The paramedian flap skin incision involves making a skin incision approximately 2-3 cm lateral to the sternal bone incision, then lifting the skin as a flap using subcutaneous tissue. The investigators aim to determine the efficacy of the paramedian flap skin incision by comparing it with the classic median skin incision, considering that this flap-style incision may result in faster wound healing and better protection against infections.

In a six-month period, 90 consecutive patients who underwent open heart surgery with classic median sternotomy in the Cardiovascular Surgery Clinic will be randomized into two groups: classic median skin incision and paramedian flap skin incision. The investigators will prospectively record data from 45 individuals in both groups and will follow them up at the first week, first month, and third month after discharge. During the follow-ups, physical examinations will be performed, wound sites and sternal bone healing processes will be evaluated, and infection status will be checked through radiologic and laboratory examinations.

Surgical Technique

Classic Median Sternotomy Skin Incision:

After the anesthesia procedures are completed in the supine position, under general anesthesia, following skin disinfection and sterile dressing, a longitudinal skin incision is made in the midline of the sternum from the jugulum to the xiphoid. Subcutaneous hemorrhages are cauterized, the periosteum is scratched in the midline with electrocautery, and a sternotomy is performed with a sternum saw, after which open heart surgery procedures are continued. In closure, after the sternum is closed, the subcutaneous tissue is first closed with the continuous suture technique, and then the skin is closed.

Para-Median Flap Skin Incision:

After the anesthesia procedures are completed in the supine position, under general anesthesia, following skin disinfection and sterile dressing, the midline of the sternum is determined. A crescent-shaped paramedian skin incision is made on the right or left side from the jugulum to the xiphoid. The subcutaneous tissue is carefully separated and opened as a flap with a dissector. Bleeding is stopped with pressure if possible, and the use of electrocautery is minimized. The periosteum is incised down to the sternal bone tissue, and the midline of the sternum is drawn with electrocautery. A sternotomy is performed, and open heart surgery procedures are continued. After the sternum is closed, the flap ends are first joined subcutaneously to ensure that the skin incision is away from the bone incision.

Data Analysis:

Demographic data of the individuals, as well as preoperative, postoperative, and follow-up data, will be recorded and analyzed using the SPSS statistical program.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective open heart surgery via median sternotomy.
* Age range: Over 18 and under 80 years of age.

Exclusion Criteria:

* Who do not accept informed consent,
* Failure to show up for necessary check-ups,
* Emergency surgery (not elective emergencies),
* Patients with exitus in the hospital in the postoperative period and during the 3-month follow-up period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who underwent open heart surgery through a classic median sternotomy at a six-month period were randomized to receive a classic median skin incision and a paramedian flap skin incision.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Determination of the effectiveness of paramedian flap skin incision technique. | 1 week, 3 month
  Observation of wound epithelization and healing process.

SECONDARY OUTCOMES:
Surgical wound infection development | 1 week, 3 month
  A sternal wound infection was defined as conditions ranging from any non-hemorrhagic discharge to a deep sternal infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)